CLINICAL TRIAL: NCT00236561
Title: A Randomized, Double-Blind, Parallel-Group, Dose-Response Study to Evaluate the Efficacy and Safety of Two Doses of Topiramate Compared to Placebo and Propranolol in the Prophylaxis of Migraine
Brief Title: A Study of the Efficacy and Safety of Two Doses of Topiramate Compared to Placebo and Propranolol in the Prevention of Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003205
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Migraine; Common Migraine; Classic Migraine; Headache
Keywords: Migraine; Common Migraine; Classic Migraine; Headache; Topiramate; Propranolol; Prophylaxis; Prevention
MeSH Terms: conditions — Migraine Disorders; Migraine without Aura; Migraine with Aura; Headache | interventions — Topiramate; Propranolol

INTERVENTIONS:
Drug: topiramate, propranolol

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of two doses of topiramate (100 and 200 mg daily) versus placebo and propranolol in the prevention of migraine. The study will also assess dose response relationship of topiramate, estimate the relative efficacy of topiramate versus propranolol in prevention of migraine, and evaluate the effect of migraine prevention with topiramate versus placebo on Health Related Quality of Life.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, multicenter study to evaluate the efficacy and safety of two doses of topiramate versus placebo and propranolol in the prevention of migraine headaches. The study consists of 4 phases: Baseline Phase (evaluation of eligibility criteria and tapering of any migraine prophylaxis medications patients are taking), Core Double-Blind Phase (patients are randomized to receive either 100 milligrams[mg]/day topiramate, 200mg/day topiramate, 160mg/day propranolol or placebo for a total of 26 weeks), Blinded Extension Phase (patients continue the same dose of medication until the sponsor terminates the study or a patient withdraws from the study), and Taper/Exit Phase (medication of patients exiting from the study is tapered over 7 weeks). The primary hypothesis is that one or two topiramate doses (100, 200 mg/day) will be superior to placebo in the prophylaxis of migraine based on the change in the monthly (28 days) migraine period rate from the prospective Baseline Phase to the Core Double-Blind Phase. Oral medication (100 milligrams[mg]/day topiramate, 200mg/day topiramate, 160mg/day propranolol, or placebo) during the 26-weeks Core Double-Blind Phase. Doses may be continued until the termination of the study or withdrawal by the patients during the Blinded Extension Phase.

ELIGIBILITY:
Inclusion Criteria:

* Medical history consistent with migraine with or without aura according to the International Headache Society (IHS) for at least 1 year prior to the study
* Between 3 to 12 migraine periods and no greater than 15 headache days (migraine and non-migraine) per month during the Baseline Phase
* No clinically significant abnormalities on neurological exams, electrocardiogram (ECG) or clinical laboratory test results at baseline
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing abstinence, or practicing an acceptable method of contraception (requires negative pregnancy test)

Exclusion Criteria:

* Patients with headaches other than migraine
* Patients with episodic tension or sinus headaches
* Onset of migraine after age of 50 years
* Patients who have failed more than two adequate regimens for migraine prophylaxis
* Patients who overuse pain medications or certain other medications

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 786 (Actual)
Dates: Start 2001-04; Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Change in the monthly (28 days) migraine period rate from the Prospective Baseline Period to the Core Double-Blind Phase.

SECONDARY OUTCOMES:
Proportion of patients responding to treatment.Change from Baseline Phase to Core Double-Blind Phase in number of monthly migraine attacks,monthly migraine days, number of days/month requiring rescue medication,and Health Related Quality of Life measures

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Diener HC, Tfelt-Hansen P, Dahlof C, Lainez MJ, Sandrini G, Wang SJ, Neto W, Vijapurkar U, Doyle A, Jacobs D; MIGR-003 Study Group. Topiramate in migraine prophylaxis--results from a placebo-controlled trial with propranolol as an active control. J Neurol. 2004 Aug;251(8):943-50. doi: 10.1007/s00415-004-0464-6. PMID 15316798